CLINICAL TRIAL: NCT04348370
Title: Bacillus Calmette-Guerin Vaccination as Defense Against SARS-CoV-2: A Randomized Controlled Trial to Protect Health Care Workers by Enhanced Trained Immune Responses
Brief Title: BCG Vaccine for Health Care Workers as Defense Against COVID 19
Acronym: BADAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Baylor College of Medicine (Other); M.D. Anderson Cancer Center (Other); Cedars-Sinai Medical Center (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0432F
Record Dates: First submitted 2020-03-30; First posted 2020-04-16 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Coronavirus; Coronavirus Infection; Coronavirus as the Cause of Diseases Classified Elsewhere
Keywords: BACILLUS CALMETTE-GUÉRIN VACCINATION; BCG Vaccine; Coronavirus; SARS-CoV-2; COVID19; COVID
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to BCG:placebo in a 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: Randomization will be done centrally and computer generated with stratification per hospital in random blocks of 2, 4 and 6. The BCG vaccine will be administered by research nurses. Participants and investigators will be blinded. The research nurse that administers the BCG vaccine or placebo will not be blinded. This research nurse will not be involved in the collection of outcome data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG Group (Experimental): FDA-approved BCG Tice strain, procured from Merck, will be used. The vaccine will be reconstituted according to the package insert. In brief, a vial containing ~1x10^8 CFU of lyophilized BCG will be reconstituted in 50 mL of saline. A single dose will consist of 0.1 mL (~2x10^5 CFU) will be administered by slow intradermal injection using a 25 gauge/ 0.5 mm syringe in the deltoid area.
  Interventions: Biological: BCG Vaccine
- Placebo Group (Placebo Comparator): A single dose will consist of 0.1 mL saline
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: BCG Vaccine — BCG vaccine will be administered by research nurses. Participants and investigators will be blinded.
  Arms: BCG Group
Biological: Placebo Vaccine — Placebo vaccine will be administered by research nurses. Participants and investigators will be blinded.
  Arms: Placebo Group

SUMMARY:
SARS-CoV-2 spreads rapidly throughout the world. A large epidemic would seriously challenge the available hospital capacity, and this would be augmented by infection of healthcare workers (HCW). Strategies to prevent infection and disease severity of HCW are, therefore, desperately needed to safeguard continuous patient care. Bacille Calmette-Guérin (BCG) is a vaccine against tuberculosis, with protective non-specific effects against other respiratory tract infections in in vitro and in vivo studies, and reported morbidity and mortality reductions as high as 70%. Furthermore, in our preliminary analysis, areas with existing BCG vaccination programs appear to have lower incidence and mortality from COVID191. The investigators hypothesize that BCG vaccination can reduce HCW infection and disease severity during the epidemic phase of SARS-CoV-2.

DETAILED DESCRIPTION:
Study design: A placebo-controlled adaptive multi-center randomized controlled trial.

Study population: High risk HCW with direct patient contacts, defined as physician assistants, respiratory therapists, nurses, physicians or other HCWs working at emergency rooms, ICUs and in locations within hospitals where COVID-infected patients are treated.

Intervention: Participants will be randomized between intradermal administration of BCG vaccine or placebo in a 1:1 ratio.

Recruitment, Randomization, treatment allocation, and blinding

A standardized, IRB approved email will be sent to department chairs describing the study. A research coordinator will reach out to interested participants via phone with the help of an IRB-approved verbal script to introduce the study, confirm eligibility and provide further instructions on how to access and sign the IRB-approved ICD via REDCap using their own electronic devices. It is important that the investigators obtain the consent via REDCAp to a) avoid direct person-to-person contact and comply with social distancing imposed recommendations, and b) minimize the waste of reconstituted BCG by allowing the research personnel to schedule vaccinations in a controlled fashion. Patient registration into the trial will happen immediately after consent has been provided and will involve entering of baseline information into an electronic data capture system (RedCap).

Once the eligibility is confirmed and the ICD signed by the participant and stored in REDCap, the research coordinator will randomize the participant and communicate the treatment assignment to the nurse administering the vaccination. The nurse will subsequently assign an appointment and communicate date and time of vaccination with the participant. All eligible participants will receive intradermal injections of BCG:placebo in a 1:1 ratio.

Both, participants and investigators will be blinded to the treatment assignments during the study. However, in case of an emergency where it is important to know the treatment received, the investigator and/or participant can reach out to the unblinded study personnel who will provide the unblinded data. All participants will receive their treatment allocation at the end of the study, after the data analysis is finalized.

Unblinded personnel will not be involved in the collection and analysis of study data other than the baseline eligibility criteria.

The end of the study is defined as the last patient's last entry in the electronic data capture system.

Informed Consent and Eligibility

The following types of procedures will be conducted as indicated below:

Medical history will be obtained from patient medical record/clinical chart. Informed Consent will be obtained to access these records. When information cannot be obtained or is not available from the patient medical record/clinical chart, it will be obtained via patient interview. Physical examination will be conducted solely to look for existing BCG vaccination scars.

Symptom evaluation will be conducted via an electronic survey administered to participants every 1-3 days.

HIV and pregnancy will be collected as self-reported information. If unknown, a urine pregnancy test will be performed.

Nasopharyngeal, oral and/ or rectal swabs will be collected for rt-PCR test for SARS-CoV2 infection if a study develops symptoms consistent with Covid-19.

If a participant does not know their PPD/IGRA status from within the last 24 months (all health care providers should have this information), an IGRA can be performed to evaluate eligibility.

Study participants have the option of donating blood via phlebotomy (for serological test for Covid-19 disease and PBMCs for immune correlates) or providing a fingerstick and dried blood spot (for serologic test for Covid-19).

Data will be collected at four time points/periods: (1) after consent, (2) at baseline, (3) during follow-up period, and (4) at study end.

Data to be collected during screening includes medical history, physical exam results, results of rt-PCR and serological test results.

Data to be collected during baseline enrollment includes eligibility confirmation, demographic information, risk factors, randomization assignment, confirmation of BCG vaccination/placebo, any immediate reactions to BCG vaccination/placebo.

Data to be collected during follow-up includes intermittent surveys about the presence of flu-like symptoms, rt-PCR test results if done, serological test results, if testing positive for Covid-19 information regarding their disease course, and disease outcome status.

THE FOLLOWING IS COLLECTED AFTER CONSENT IS OBTAINED:

Date of signed Informed Consent Form

Role in hospital

Department in hospital

rt-PCR test for SARS-CoV2 result

Serological test for Covid-19 result

Number of BCG scars (by visual/physical examination)

Medical history*

Previous PPD and IGRA test results

History of TB disease

History of previous HIV testing

Urine Pregnancy test result (if applicable)

Plans of pregnancy in 30 days

Plan to stop working in 3 months/ leave facility in 6 months

Current diabetes mellitus

Current chronic kidney disease

Currently taking immunosuppressive drugs

Living with someone with HIV, immunocompromised, taking immunosuppressive drug

Chemotherapy in past 3 months

History of organ/bone marrow transplant

Access to smartphone

BASELINE DATA COLLECTION/PROCEDURES

The following procedures will be conducted and data collected as indicated below:

A questionnaire to obtain information about age, sex, demographic information, who they live with, smoking status, any current medications they are on, and other comorbidities

Participants will then be randomized to either receive a single dose of BCG vaccination or placebo.

BCG vaccination or placebo will be administered.

Eligibility screening data will carry forward into the trial.

The following additional data points will be collected:

Age

Sex

Race

Ethnicity

Nationality

Who they live with

Height

Weight

Smoking status/tobacco use

Alcohol use

Current list of medications

Current list of comorbidities

History of diabetes mellitus

History of hypertension

History of stroke

History of kidney disease

History of COPD

Randomization assignment

BCG/placebo administered

FOLLOW-UP PROCEDURES AND DATA COLLECTION:

Participants will be followed to assess whether they get infected with SARS-CoV2:

Participants will complete intermittent surveys via an electronic system every 1-3 days to assess the presence of any flu-like symptom, including sore throat, fever, headache, malaise, and cough. Note that this is part of routine surveillance for Covid-19 in health workers at the United States site. Consent forms will ask for consent to access this survey information.

Any positive response on the survey will trigger a nasopharyngeal, oral and/ or rectal swab to be collected to test for Covid-19 via rt-PCR

All participants, regardless of survey responses, will have serology for Covid-19 tested at 4 week intervals during the follow-up period (6 months)

If a participant completes the follow-up period and does not test positive for disease, their study participation is complete

If a participant does test positive for disease, their disease status will be ascertained for up to two months or until an outcome is available through one of the following mechanisms: (1) an electronic survey if they are not admitted to the hospital, including questions about the number of days they are ill, daily fever, and other symptoms; or (2) (2) if they are admitted to the hospital, ordinal outcomes for disease severity will be extracted from the hospital¿s electronic medical records system.

During the first week of follow-up, all participants will actively be asked about any adverse events; thereafter, participants will report unsolicited AEs through the electronic survey. Vaccine related adverse events will be graded using the FDA guidance (https://www.fda.gov/media/73679/download) and noted using WHO-recommended Adverse event following Immunization forms (AEFI; https://vaccine-safety-training.org/classification-of-aefis.html).

Participants will have the option of donating 12 mL of blood for plasma (serology) and PBMCs for secondary analysis of immune correlates and for future analysis based on covid19-specific IgM and IgG. If they do not donate 12mL of blood, a fingerstick will be required for baseline COVID19 serology.

Dried Blood Spot (DBS): all participants are HCWs and will self-collect DBS samples at week 4, 8, 12, 16, 20 and 24. Envelopes to store the DBS are provided upon enrollment and can be dropped off at work and picked up by study coordinators to minimize HCW distractions.

COVID specific RNA is found in stool for ~21 days when an individual develops infection (https://doi.org/10.1038/s41586-020-2196-x). Participants will have the option of collecting stool swabs monthly if they are asymptomatic or weekly if they develop symptoms. Nucleic acid testing will be performed in retrospect to support secondary objectives.

If participants develop symptoms consistent with COVD19, will be PCR tested for COVID19. They will be given the option of donating 12 mL of blood for plasma and PBMCs 2 weeks after symptoms resolve.

Week 12 (+/- 2 Weeks), participants will be given the option to donate 12 mL of blood for plasma and PBMCs for secondary analysis of immune correlates and for future secondary analysis based on covid-specific IgM and IgG.

Week 24 (+/- 2 Weeks), participants will be given the option to donate 12 mL of blood for plasma and

PBMCs for secondary analysis of immune correlates and for future secondary analysis based on covid-specific IgM and IgG.

Except for the administration of BCG vaccine or placebo and the above mentioned DBS and phlebotomy, participants will undergo no invasive procedures for study purposes.

The following data points will be collected during the follow-up period AND AT

END OF STUDY TIMEPOINT:

Sore throat (collected at multiple time points)

Fever (collected at multiple time points)

Headache (collected at multiple time points)

Malaise (collected at multiple time points)

Cough (collected at multiple time points)

rt-PCR test for SARS-CoV2 result (as indicated)

Serological test for Covid-19 result (every 2 weeks)

Number of days ill

Daily fever

Other Covid-19 symptoms

Admitted to hospital

Required oxygen

Treated in intensive care

Required ventilation

Death

Severe pneumonia

Respiratory failure

Acute respiratory distress syndrome

Sepsis

Septic shock

*Already being collected as part of routine surveillance of health care workers. Will request access to this information in Informed Consent Form.

Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons. Participants who received placebo will be unblinded at the end of the study and pending a recommendation by the DSMB, they will be offered the option of receiving the BCG intervention.

A participant will only be replaced in case of withdrawal before the administration of BCG vaccine/placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Male or female
* Hospital personnel taking care for patients with known or suspected SARS-CoV-2 infection and providing, on average, at least 25 hours per week of direct patient care

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious adverse events to prior BCG administration
* Known active or latent Mycobacterium tuberculosis or with another mycobacterial species. A history with- or a suspicion of M. tuberculosis infection.
* Fever (>38 C) within the past 24 hours
* Age > 75 years
* Pregnancy or planning pregnancy within 30 days of study enrollment
* Breastfeeding
* Suspicion of active viral or bacterial infection
* Any Immunocompromised subjects. This exclusion category comprises: a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) subjects with known neutropenic with less than 1500 neutrophils/mm3; c) subjects with solid organ transplantation; d) subjects with bone marrow transplantation; e) subjects under chemotherapy; f) subjects with primary immunodeficiency; g) known severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any anti-cytokine therapies. i) treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months
* Living with someone who is immunosuppressed or taking immunosuppressive drugs
* Previous documented infection with COVID19
* Active solid or non-solid malignancy or lymphoma within the prior two years
* Direct involvement in the design or the execution of the study
* Expected absence from work of ≥4 of the following 12 weeks due to any reason (holidays, maternity leave, retirement, planned surgery etc)
* Not in possession of a smartphone
* Inability to keep the vaccine site covered in the case of a draining pustule.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Cirillo, PhD, Principal Investigator — Texas A&M University; Andrew DiNardo, MD, Principal Investigator — Baylor College of Medicine; Ashish M Kamat, MD, Principal Investigator — M.D. Anderson Cancer Center; Moshe Arditi, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Texas A&M Family Care Clinic, Bryan, Texas
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Harris Health System - Ben Taub Hospital, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Chang D, Xu H, Rebaza A, Sharma L, Dela Cruz CS. Protecting health-care workers from subclinical coronavirus infection. Lancet Respir Med. 2020 Mar;8(3):e13. doi: 10.1016/S2213-2600(20)30066-7. Epub 2020 Feb 13. No abstract available. PMID 32061333
- [Background] Zhang J, Zhou L, Yang Y, Peng W, Wang W, Chen X. Therapeutic and triage strategies for 2019 novel coronavirus disease in fever clinics. Lancet Respir Med. 2020 Mar;8(3):e11-e12. doi: 10.1016/S2213-2600(20)30071-0. Epub 2020 Feb 13. No abstract available. PMID 32061335
- [Background] Benn CS, Netea MG, Selin LK, Aaby P. A small jab - a big effect: nonspecific immunomodulation by vaccines. Trends Immunol. 2013 Sep;34(9):431-9. doi: 10.1016/j.it.2013.04.004. Epub 2013 May 14. PMID 23680130
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537
- [Background] Kristensen I, Aaby P, Jensen H. Routine vaccinations and child survival: follow up study in Guinea-Bissau, West Africa. BMJ. 2000 Dec 9;321(7274):1435-8. doi: 10.1136/bmj.321.7274.1435. PMID 11110734
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Nemes E, Geldenhuys H, Rozot V, Rutkowski KT, Ratangee F, Bilek N, Mabwe S, Makhethe L, Erasmus M, Toefy A, Mulenga H, Hanekom WA, Self SG, Bekker LG, Ryall R, Gurunathan S, DiazGranados CA, Andersen P, Kromann I, Evans T, Ellis RD, Landry B, Hokey DA, Hopkins R, Ginsberg AM, Scriba TJ, Hatherill M; C-040-404 Study Team. Prevention of M. tuberculosis Infection with H4:IC31 Vaccine or BCG Revaccination. N Engl J Med. 2018 Jul 12;379(2):138-149. doi: 10.1056/NEJMoa1714021. PMID 29996082
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Han RF, Pan JG. Can intravesical bacillus Calmette-Guerin reduce recurrence in patients with superficial bladder cancer? A meta-analysis of randomized trials. Urology. 2006 Jun;67(6):1216-23. doi: 10.1016/j.urology.2005.12.014. PMID 16765182
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Spencer JC, Ganguly R, Waldman RH. Nonspecific protection of mice against influenza virus infection by local or systemic immunization with Bacille Calmette-Guerin. J Infect Dis. 1977 Aug;136(2):171-5. doi: 10.1093/infdis/136.2.171. PMID 894076
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Joosten LA, Ifrim DC, Saeed S, Jacobs C, van Loenhout J, de Jong D, Stunnenberg HG, Xavier RJ, van der Meer JW, van Crevel R, Netea MG. Bacille Calmette-Guerin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A. 2012 Oct 23;109(43):17537-42. doi: 10.1073/pnas.1202870109. Epub 2012 Sep 17. PMID 22988082
- [Background] Kleinnijenhuis J, Quintin J, Preijers F, Benn CS, Joosten LA, Jacobs C, van Loenhout J, Xavier RJ, Aaby P, van der Meer JW, van Crevel R, Netea MG. Long-lasting effects of BCG vaccination on both heterologous Th1/Th17 responses and innate trained immunity. J Innate Immun. 2014;6(2):152-8. doi: 10.1159/000355628. Epub 2013 Oct 30. PMID 24192057
- [Background] Leentjens J, Kox M, Stokman R, Gerretsen J, Diavatopoulos DA, van Crevel R, Rimmelzwaan GF, Pickkers P, Netea MG. BCG Vaccination Enhances the Immunogenicity of Subsequent Influenza Vaccination in Healthy Volunteers: A Randomized, Placebo-Controlled Pilot Study. J Infect Dis. 2015 Dec 15;212(12):1930-8. doi: 10.1093/infdis/jiv332. Epub 2015 Jun 12. PMID 26071565
- [Background] Arts RJ, Blok BA, Aaby P, Joosten LA, de Jong D, van der Meer JW, Benn CS, van Crevel R, Netea MG. Long-term in vitro and in vivo effects of gamma-irradiated BCG on innate and adaptive immunity. J Leukoc Biol. 2015 Dec;98(6):995-1001. doi: 10.1189/jlb.4MA0215-059R. Epub 2015 Jun 16. PMID 26082519
- [Background] Cheng SC, Quintin J, Cramer RA, Shepardson KM, Saeed S, Kumar V, Giamarellos-Bourboulis EJ, Martens JH, Rao NA, Aghajanirefah A, Manjeri GR, Li Y, Ifrim DC, Arts RJ, van der Veer BM, Deen PM, Logie C, O'Neill LA, Willems P, van de Veerdonk FL, van der Meer JW, Ng A, Joosten LA, Wijmenga C, Stunnenberg HG, Xavier RJ, Netea MG. mTOR- and HIF-1alpha-mediated aerobic glycolysis as metabolic basis for trained immunity. Science. 2014 Sep 26;345(6204):1250684. doi: 10.1126/science.1250684. PMID 25258083
- [Background] Shivayogi P. Vulnerable population and methods for their safeguard. Perspect Clin Res. 2013 Jan;4(1):53-7. doi: 10.4103/2229-3485.106389. No abstract available. PMID 23533983
- [Derived] DiNardo AR, Arditi M, Kamat AM, Koster KJ, Carrero S, Nishiguchi T, Lebedev M, Benjamin AB, Avalos P, Lozano M, Moule MG, McCune B, Herron B, Ladki M, Sheikh D, Spears M, Herrejon IA, Dodge C, Kumar S, Hutchison RW, Ofili TU, Opperman LA, Bernard JA, Lerner SP, Udeani G, Neal G, Netea MG, Cirillo JD. Bacillus Calmette-Guerin vaccination as defense against SARS-CoV-2 (BADAS): a randomized controlled trial to protect healthcare workers in the USA by enhanced trained immune responses. Trials. 2023 Oct 4;24(1):636. doi: 10.1186/s13063-023-07662-w. PMID 37794431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCG Group | Placebo Group
Started | 334 | 325
Completed | 263 | 266
Not Completed | 71 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCG Group | Placebo Group | Total
Number analyzed (Participants) | 334 | 325 | 659
Age, Continuous [Median (Standard Deviation); unit: years] | 47.01 (12.3) | 46.6 (12.4) | 46.81 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 215 | 222 | 437
  Male | 119 | 103 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 59 | 102
  Not Hispanic or Latino | 291 | 266 | 557
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 37 | 32 | 69
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 5 | 9 | 14
  White | 276 | 266 | 542
  More than one race | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 334 | 325 | 659
Prior BCG [Number; unit: participants] | 28 | 35 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of New COVID 19 Infections
Description: The primary outcome measure is development of COVID19 infection. This will be reported as the number of individuals receiving the intervention who are PCR-positive or seroconvert, defined as number of new cases during the 6 month time period
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | BCG Group | Placebo Group
Number analyzed (Participants) | 263 | 266
Participants | 25 | 21

2. Secondary Outcome: Disease Severity
Description: The secondary outcome measure is disease severity calculated using the Covid Severity Scale Scoring of 0 -10. A score of 10 is worse and a score of 0 is best. Disease severity score will be based on the level of care required for individuals who test positive for COVID19 as follows: non-hospital-based care; patient hospitalized but no oxygen required; hospitalized and oxygen required; patient treated in intensive care and/or on mechanical ventilation; patient died. Additional WHO criteria for severity include severe pneumonia, respiratory failure, acute respiratory distress syndrome, sepsis and septic shock.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | BCG Group | Placebo Group
Number analyzed (Participants) | 25 | 21
score on a scale | 2 [2 to 2] | 2 [2 to 2]

ADVERSE EVENTS:
Time Frame: Data were collected during the 6 months of the study plus a 6 month optional followup period for disease outcome.
Description: Participants reported unsolicited AEs through the electronic survey.
Arm/Group | BCG Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/266
Serious Adverse Events (participants affected / at risk) | 1/263 | 0/266
Other Adverse Events (participants affected / at risk) | 75/263 | 73/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCG Group (N=263) | Placebo Group (N=266)
Dental caries (Injury, poisoning and procedural complications) | 1 | 0 — Participant broke tooth while eating. It was determined the tooth could not be salvaged and was removed. An implant would be required. The patient had the procedure to start the implant process. Patient states they have had no further issues.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCG Group (N=263) | Placebo Group (N=266)
Cough, headache, myalgias (General disorders) | 75 | 73 — Subjects displayed one of the following symptoms, either a cough, headache or myalgias. In most cases not displayed together.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-31): https://cdn.clinicaltrials.gov/large-docs/70/NCT04348370/Prot_SAP_000.pdf